CLINICAL TRIAL: NCT02219126
Title: Effect of Homogenization and Pasteurization of Milk on the Stomach Problems in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, PhD, Adjunct professor, University of Turku
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MILK
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Unidentified Stomach Discomfort Following Dairy Consumption
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homogenized and pasteurized milk (Experimental): Milk that has undergone homogenization ans pasteurization treatment
  Interventions: Other: Dietary intervention
- Nonhomogenized and nonpasteurized milk (Experimental): Unhomogenized and unpasteurized milk (raw milk)
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention

SUMMARY:
This study aims to investigate differences in digestion rates and stomach problems caused by pasteurized and homogenized milk compared with raw milk in healthy adults by ingestible capsule that measures pH and pressure, diary of symptoms, blood glucose and triacylglycerol levels and plasma cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

* Homogenized and pasteurized milk causes stomach problems (self-reported)
* unhomogenized and unpasteurized milk does not cause stomach problems (self-reported)
* age 18-65
* BMI 18,5 - 30
* hemoglobin under normal range
* fasting plasma alanine aminotransferase ALAT < 60 U/l (normal liver function)
* fasting plasma thyroid-stimulating hormone (TSH) 0.4 - 4.5 mU/l (normal thyroid function)
* fasting plasma creatinine < 118 umol/l (normal kidney function)

Exclusion Criteria:

* pace maker
* Crohn's disease or other disease of the intestinal tract
* intestinal operation within the last 3 months
* difficult dysphagia
* smoking
* constipation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Pressure in the intestinal tract | Day 0 - Day 5
  Pressure in the intestinal tract as measured by ingestible Smart Pill -capsule.
Gastrointestinal symptoms (self-reported) | Day 0 - Day 5
  Gastrointestinal symptoms (self-reported) as measured by a questionnaire. The questionnaire is devided into seven types of stomach discomfort, and also includes a possibility to describe a stomach discomfort outside these seven given alternatives. The severity of the symptoms is self-reported on a three-step scale.

SECONDARY OUTCOMES:
Plasma triacylglycerols | 20min, 40min, 60min, 120min, 180min, 240min
Plasma glucose | 20min, 40min, 60min, 90min, 120min, 180min, 240min
Plasma triacylglycerols | 20min, 40min, 60min, 90min, 120min, 180min, 240min
Plasma insulin | 20min, 40min, 60min, 90min, 120min, 180min, 240min

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa M Linderborg, PhD, Principal Investigator — University of Turku
Locations (1):
- Department of Biochemistry University of Turku, Turku, Finland